CLINICAL TRIAL: NCT00680706
Title: Targeting Myocardial Energy Metabolism for the Treatment of Acute Heart Failure: The Effect of Thiamine on Biochemical, Electrocardiographic and Respiratory Parameters in Hospitalized Patients.
Brief Title: Thiamine and Acute Decompensated Heart Failure: Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Howard Smithline, Chief, Emergency Medicine Research, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-059
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure; Diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus | interventions — Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thiamine (Experimental): Receives thiamine
  Interventions: Drug: Thiamine
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Thiamine — Thiamine (100 mg) in 50 ml D5W, x 2.
  Other Names: Vitamin B1
  Arms: Thiamine
Drug: Placebo — D5W (50 ml)
  Arms: Control

SUMMARY:
Heart failure remains an increasing cause of morbidity and mortality in the United States even in the face of recent advances in the treatment of cardiovascular disease. There is an urgent need to reevaluate the treatment of heart failure. Shifting substrate utilization used in energy metabolism from fatty acids to glucose is beneficial to the heart presumably by increasing the efficiency of ATP production. Several new drugs for the treatment of cardiac ischemia work by this mechanism. There is increasing evidence that patients with heart failure may also benefit by the same type of intervention. Patients with heart failure are known to have low serum thiamine levels because of poor dietary intake and increased urinary excretion. Inadequate thiamine will deleteriously shift substrate utilization from glucose to fatty acids.

We hypothesize that thiamine supplementation will be beneficial for patients with heart failure by increasing glucose and decreasing fatty acid utilization. This will be initially tested in a pilot double-blinded placebo controlled study of thiamine supplementation in diabetic and non-diabetic patients presenting to the emergency department with acute decompensated heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. History of heart failure on a loop diuretic.
2. Worsening dyspnea over the past 24 hours.
3. Currently dyspneic sitting or supine, on or off oxygen.
4. Radiographic cephalization of vessels. This criteria is not needed if the patient has no other reason for being dyspneic after being evaluated in the emergency department.
5. Elevated NT pro-BNP (>450).
6. Able to communicate in English or Spanish.
7. Able and willing to provide informed consent.
8. Age > 18 years.
9. A primary admitting diagnosis of acute decompensated heart failure.

Exclusion Criteria:

1. Renal failure on dialysis.
2. Severe valvular disease.
3. EKG criteria for acute myocardial infarction (ST segment elevation > 1mm on two contiguous leads).
4. Initial troponin elevated.
5. Ventricular arrhythmia (ventricular tachycardia or fibrillation).
6. Supraventricular arrhythmia (atrial fibrillation / flutter) with a ventricular rate >120 beats per minute.
7. Taking a daily thiamine supplementation (any multivitamin or specific thiamine supplementation within the past 2 weeks. Fortified foods, such as cereals, are acceptable
8. Taking a daily fatty acid supplement.
9. Pregnancy as determined by standard serum or urine b-HCG assay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-01; Primary Completion 2010-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Smithline, MD, Principal Investigator — Baystate Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts

REFERENCES:
- [Derived] Smithline HA, Donnino M, Blank FSJ, Barus R, Coute RA, Knee AB, Visintainer P. Supplemental thiamine for the treatment of acute heart failure syndrome: a randomized controlled trial. BMC Complement Altern Med. 2019 May 6;19(1):96. doi: 10.1186/s12906-019-2506-8. PMID 31060559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: January 2008 to February 2010 Location: Emergency Department
Pre-assignment Details: One subject was dropped by the PI after consent but before randomization because the subject did not meet the inclusion/exclusion criteria.
Groups:
- Thiamine: Receives thiamine, 100 mg intravenously at baseline (time 0-hour) and again at time 24-hour.
- Control: Receives placebo
Period: Overall Study
Arm/Group | Thiamine | Control
Started | 70 | 60
Completed | 63 | 55
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiamine | Control | Total
Number analyzed (Participants) | 70 | 60 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 73 (13) | 73 (13) | 73 (13)
Sex/Gender, Customized [Number; unit: participants]
  Male | 34 | 33 | 67
  Female | 33 | 27 | 60
  Unknown | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of Thiamine Supplementation on Dyspnea
Description: Sitting Upright on Oxygen. Measured using a 10-centimeter visual analog scale (VAS). Measures are in units of millimeters (mm). A smaller number should be interpreted as a less dyspnea. A larger number should be interpreted as a more dyspnea. Less dyspnea is a better clinical outcome than more dyspnea.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: mm
Groups:
- Control: Placebo
Arm/Group | Control | Thiamine
Number analyzed (Participants) | 55 | 63
mm | 34 [28 to 40] | 32 [26 to 37]

2. Primary Outcome: Effect of Thiamine Supplementation on Dyspnea
Description: as for outcome 1
Time Frame: 8-Hour
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Control | Thiamine
Number analyzed (Participants) | 55 | 63
mm | 19 [12 to 26] | 28 [22 to 34]

ADVERSE EVENTS:
Arm/Group | Thiamine | Control
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/55
Other Adverse Events (participants affected / at risk) | 0/63 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes